CLINICAL TRIAL: NCT04482634
Title: Is Tele-rehabilitation Superior to Home Exercise Program in the Pulmonary Rehabilitation of the Patients With COVID-19 With Post-intensive Care Syndrome? A Randomized Controlled Trial
Brief Title: Tele-rehabilitation Versus Home Exercise Program in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.219.IRB1.069
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Rehabilitation; COVID-19
Keywords: pulmonary rehabilitation; COVID-19; pulmonary exercise; post-intensive care syndrome
MeSH Terms: conditions — COVID-19; postintensive care syndrome

STUDY DESIGN:
Intervention Model Description: There will be two groups. The first group will perform the exercises at their home under remote supervision (tele-rehabilitation group) and the second group will perform the exercises at their home on their own (home exercise group)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation group (Active Comparator): This group will perform the exercises at their home under remote supervision of a physiotherapist via internet connection.
  Interventions: Other: Remote controlled exercise
- Home exercise group (Active Comparator): This group will perform the exercises at their home on their own, the first exercise program will be given at hospital and the patients will be followed up regular weekly by phone call.
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Remote controlled exercise — Breathing, aerobic, posture, stretching, upper and lower extremity strengthening exercises.
  Arms: Tele-rehabilitation group
Other: Home exercise — Breathing, aerobic, posture, stretching, upper and lower extremity strengthening exercises.
  Arms: Home exercise group

SUMMARY:
The aim of the study is to investigate the potential effects of face-to-face supervised tele-rehabilitation to home exercise program on walking speed, handgrip strength, muscle endurance, quality of life, physical activity level and perceived respiratory disability in COVID-19 patients who hospitalized in ICU due to ARDS and discharged from hospital.

DETAILED DESCRIPTION:
COVID-19 could cause respiratory distress in a minority of cases and requires intensive care and mechanical ventilation. When patients recover and are discharged from hospital, physical, cognitive and emotional complications known as post-intensive care syndrome is seen in the majority of patients and requires rehabilitation.

Pulmonary rehabilitation is a comprehensive intervention consists of assessment of patient, exercise training and education in order to improve physical and psychological condition of people with chronic respiratory disease.

The patients with COVID-19 with post-intensive care syndrome will be randomized two groups: Tele-rehabilitation group and home exercise group. There will not be a non-exercising control group due to the ethical issues. The exercise program of both groups will be prescribed by a physiatrist based on the physical examination and the functional capacity of the patients.

Tele-rehabilitation group will perform the exercise program 3 days/week for 10 weeks. One session will include aerobic, flexibility and strengthening exercises for lower and upper extremity and breathing exercise.

The trainings will start with low-intensity exercises and intensity and duration of the exercises will progress according to the condition of the patient.

Intensity of the exercises will be monitored by Borg scale based on dyspnea and exertion symptoms during the sessions.

Home exercise group will perform the exercises at their home on their own, 3 days/week for 10 weeks. The patients will be trained about the individualised exercise program as the first session provided at the hospital. The physiotherapist will call the patients weekly, modifications in the exercise program will be made according to the patient's reports.

Outcomes will be measured at baseline, within 1 week of completion the program, 6th months and 12th months following the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* To be older than 18 years
* To be discharged from ICU with a diagnosis of ARDS or severe pneumonia due to COVID-19
* To have ability to walk independently

Exclusion Criteria:

* To have dementia or cognitive impairment, symptomatic psychiatric illness, hearing or visual impairment that might interfere to follow the instructions
* To have a severe co-morbidity that exercise is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 12 months
  This is a field test evaluating submaximal aerobic capacity. The individuals are asked to walk as far as possible in a 30-meter corridor in 6 minutes. The technical standards are defined by European Respiratory Society and American Thoracic Society. Six-minute walking distance will be recorded. Higher walking distance shows better outcome. Minimal clinical difference is 20-30 meter in patients surviving acute respiratory distress syndrome

SECONDARY OUTCOMES:
Short form - 36 | 12 months
  Short form - 36 measures health related quality of life. It is a self-reported survey that evaluates individual health status with eight parameters consisting of physical function, pain, role limitations attributed to physical problems, role limitations attributed to emotional problems, mental health, social functioning, energy/ vitality, general health perception. There is not a summary score, each section is scored between 0-100, 0 indicates the worst condition, 100 indicates the best.
Chair- stand test | 12 months
  Chair stand test will be used to evaluate strength and endurance of lower limbs. Patients will be asked to sit on a chair by crossing their hands over their chest and sit five times consecutively as fast as possible. The test will be started in the sitting position and terminated at the last standing position and the time will be recorded. The test will be carried out 2 times and the best grade obtained will be recorded
Timed up and go test | 12 months
  To assess physical function/performance, timed up and go test will be performed. It is an objective, reliable and simple test to evaluate balance and functional movement. The patient will be asked to get up from a chair, walk 3 m, turn around, walk back and sit on the chair again. The time will be recorded in seconds. The test will be started and ended when the patient sit on the chair with back supported. It predicts mortality.
St. George's Respiratory Questionnaire | 12 months
  St. George's Respiratory Questionnaire is a 50-item questionnaire with 76 weighted responses that is developed to measure health status/ quality of life in patients with airway diseases. It consists of 3 sections; symptoms (8 item), activity (16 item) and impact of the disease (26 item). Each of the 3 sections is scored separately and a summary total score is calculated using weights attached to each item in the range 0 to 100. 0 indicates best possible health status and 100 indicates worst possible health status. A minimum change in score of 4 units was established as clinically relevant. Turkish reliability of the questionnaire is exist.
The COPD Assessment Test | 12 months
  The COPD Assessment Test evaluates 8 parameters for measuring the impact of COPD on a patient's life and how changes over time. It provides a scoring range of 0-40, higher score indicates worst health. Turkish validity and reliability of the test is exist.
Medical Research Council Dyspnea Scale | 12 months
  The Medical Research Council Dyspnea Scale is a simple method measuring perceived respiratory disability of COPD patients. It consists of 5 items from 0 to 4. 0 indicates normal, 4 indicates worst.
Hand grip strength | 12 months
  Hand grip strength is an indicator of overall muscle strength that predicts mortality in older patients and correlates with 6 minute walk distance in subjects with COPD exacerbation. Handgrip strength will be measured using a handheld dynamometer (JAMAR Plus+ electronic dynamometer, part number: 563213, serial number: 2019070814) according to the instructions of the American Society of Hand Therapists. Patients will be seated placing their arms by their sides with the elbow flexed to 90°, the forearm mid-prone, and the wrist in neutral position. Patients will be asked to grip the dynamometer with maximally to measure maximal grip strength (in kg) for the dominant hand with standard verbal encouragement. Three trials will be performed with a 30 sec rest between trials and the highest value will be recorded. The cut-off values of grip strength are 28.6 kg in men and 16.4 kg in women.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Held N, Moss M. Optimizing Post-Intensive Care Unit Rehabilitation. Turk Thorac J. 2019 Apr 1;20(2):147-152. doi: 10.5152/TurkThoracJ.2018.18172. Print 2019 Apr. PMID 30958989
- [Result] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Result] Lau HM, Ng GY, Jones AY, Lee EW, Siu EH, Hui DS. A randomised controlled trial of the effectiveness of an exercise training program in patients recovering from severe acute respiratory syndrome. Aust J Physiother. 2005;51(4):213-9. doi: 10.1016/s0004-9514(05)70002-7. PMID 16321128
- [Result] Bourne S, DeVos R, North M, Chauhan A, Green B, Brown T, Cornelius V, Wilkinson T. Online versus face-to-face pulmonary rehabilitation for patients with chronic obstructive pulmonary disease: randomised controlled trial. BMJ Open. 2017 Jul 17;7(7):e014580. doi: 10.1136/bmjopen-2016-014580. PMID 28716786
- [Result] Turan Z, Ozyemisci Taskiran O, Erden Z, Kokturk N, Kaymak Karatas G. Does hand grip strength decrease in chronic obstructive pulmonary disease exacerbation? A cross-sectional study. Turk J Med Sci. 2019 Jun 18;49(3):802-808. doi: 10.3906/sag-1811-22. PMID 31190519
- [Result] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Result] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Result] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Result] Bergland A, Jorgensen L, Emaus N, Strand BH. Mobility as a predictor of all-cause mortality in older men and women: 11.8 year follow-up in the Tromso study. BMC Health Serv Res. 2017 Jan 10;17(1):22. doi: 10.1186/s12913-016-1950-0. PMID 28068995
- [Result] Beaudart C, McCloskey E, Bruyere O, Cesari M, Rolland Y, Rizzoli R, Araujo de Carvalho I, Amuthavalli Thiyagarajan J, Bautmans I, Bertiere MC, Brandi ML, Al-Daghri NM, Burlet N, Cavalier E, Cerreta F, Cherubini A, Fielding R, Gielen E, Landi F, Petermans J, Reginster JY, Visser M, Kanis J, Cooper C. Sarcopenia in daily practice: assessment and management. BMC Geriatr. 2016 Oct 5;16(1):170. doi: 10.1186/s12877-016-0349-4. PMID 27716195